CLINICAL TRIAL: NCT06879717
Title: A Phase I/IIa Study of Roginolisib in Combination With Dostarlimab With or Without Docetaxel in Patients With Advanced Non-squamous NSCLC Who Have Progressed on Standard of Care Immune Checkpoint Therapy and Platinum Doublet Chemotherapy or Standard Immunotherapy Without Chemotherapy (PULMO-1)
Brief Title: A Study of Roginolisib (IOA-244) in Combination With Dostarlimab With or Without Docetaxel in Metastatic Non Small-cell Lung Cancer (NSCLC) Patients
Acronym: PULMO-01
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: iOnctura (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IOA-244-202; 2024-517741-14 (EudraCT Number)
Record Dates: First submitted 2025-03-05; First posted 2025-03-17 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer (NSCLC); Advanced Non Squamous NSCLC
Keywords: Advanced non-squamous Non Small Cell Lung Cancer
MeSH Terms: interventions — dostarlimab; Docetaxel

STUDY DESIGN:
Intervention Model Description: Randomised, parallel-arm, comparator controlled, open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Roginolisib + dostarlimab + docetaxel (Experimental): IOA-244 80 mg (corresponding to 72 mg roginolisib) once daily oral dosing on a 21-day cycle. Dostarlimab: 500 mg administered as IV infusion over 30 minutes on Day 1 of every 21-day cycle to a maximum of 35 cycles. Docetaxel: 75 mg/m2 administered over 1 hour as IV infusion on Day 1 of every 21-day cycle.
  Interventions: Drug: roginolisib; Drug: Dostarlimab; Drug: Docetaxel
- Arm 2: Roginolisib + dostarlimab (Experimental): IOA-244 80 mg (corresponding to 72 mg roginolisib) once daily oral dosing on a 21-day cycle. Dostarlimab: 500 mg administered as IV infusion over 30 minutes on Day 1 of every 21-day cycle to a maximum of 35 cycles.
  Interventions: Drug: roginolisib; Drug: Dostarlimab
- Arm 3: Dostarlimab + docetaxel (Active Comparator): Dostarlimab: 500 mg administered as IV infusion over 30 minutes on Day 1 of every 21-day cycle to a maximum of 35 cycles. Docetaxel: 75 mg/m2 administered over 1 hour as IV infusion on Day 1 of every 21-day cycle.
  Interventions: Drug: Dostarlimab; Drug: Docetaxel

INTERVENTIONS:
Drug: roginolisib — tablet, 40mg tablet strength
  Arms: Arm 1: Roginolisib + dostarlimab + docetaxel; Arm 2: Roginolisib + dostarlimab
Drug: Dostarlimab — 500 mg administered as IV infusion
Drug: Docetaxel — 75 mg/m2 administered over 1 hour as IV infusion
  Arms: Arm 1: Roginolisib + dostarlimab + docetaxel; Arm 3: Dostarlimab + docetaxel

SUMMARY:
The goal of this clinical trial is to learn how roginolisib works in combination with dostarlimab with or without docetaxel in adult patients with advanced non small-cell lung cancer. The main questions it aims to answer are:

To compare across the treatment arms the proportion of patients with a reduction in Treg cells To evaluate the safety and tolerability of roginolisib plus dostarlimab, with or without docetaxel

DETAILED DESCRIPTION:
A Phase I/IIa open-label, randomised study of oral roginolisib (IOA-244 [roginolisib hemi-fumarate]) in combination with dostarlimab with or without docetaxel in Advanced Non small-cell lung cancer (NSCLC) patients.

This study will enrol approximately 45 male and female patients aged over 18 years with advanced NSLCL who have process on standard of care immune checkpoint therapy and platinum doublet chemotherapy or standard immunotherapy without chemotherapy. The disease must be measurable (i.e., at least 1 measurable lesion) as per RECIST v1.1 by Computerised Tomography (CT) scan or Magnetic Resonance Imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age inclusive, at the time of signing the informed consent.
2. Capable of giving signed informed consent, which includes compliance with the requirements of this protocol.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
4. Histologically or cytologically confirmed stage IIIb/IV or recurrent non-squamous NSCLC.
5. Have measurable disease per RECIST v1.1 as determined by the investigator. Tumour lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
6. Documented radiographic disease progression on or after prior anti-PD(L)1 therapy and platinum chemotherapy or after standard immunotherapy without chemotherapy in accordance with standard of care.
7. Male or female patients of child-bearing potential must be willing to use highly effective forms of contraception (refer to APPENDIX 3 for details on highly effective methods of contraception and definitions of women of childbearing potential [WOCBP]and of fertile men):

   1. Women of childbearing potential (WOCBP) must have a negative serum test as per local guidelines during screening and EOT and agree to have regular urine pregnancy testing throughout the study. WOCBP must agree to use a highly effective method of contraception and refrain from donating eggs throughout the study and until 4 months after last dose of IMP;
   2. Male patients must agree to use barrier method of contraception [condom plus spermicide] from screening through Safety Follow-up visit, at least 1 month after the last dose of IMP. Men should refrain from donating sperm from the day of first dose of IMP, throughout the study and until 3 months after last dose of IMP. Men with partners of child-bearing potential must also be willing to ensure that their partner uses a highly effective method of contraception for the same duration. Men with pregnant or lactating partners should be advised to use barrier method contraception (e.g., condom plus spermicidal gel) to prevent exposure to the foetus or neonate.

Exclusion Criteria:

1. Inability to swallow food or any condition of the upper gastrointestinal tract that precludes administration of oral medications.
2. Histologically or cytologically confirmed squamous NSCLC.
3. Previously treated with dostarlimab or docetaxel.
4. Have prior significant medical history and AEs:

   1. History of a prior Grade 3 or 4 immune-related AE (irAE) or any grade ocular irAE from prior immunotherapy which did not respond to corticosteroid therapy or resolved with treatment interruptions and returned to at least Grade 1; immunemediated severe neurologic events of any grade (e.g., myasthenic syndrome/myasthenia gravis, encephalitis, Guillain-Barré Syndrome, or transverse myelitis), exfoliative dermatitis of any grade (SJS, TENS, or DRESS syndrome), or myocarditis of any grade.
   2. Have not recovered from toxic effect(s) of prior therapy to ≤ Grade 1, other than alopecia or fatigue or neuropathy which must be ≤ Grade 2.
   3. Active autoimmune process (e.g., rheumatoid arthritis, moderate or severe psoriasis, multiple sclerosis, inflammatory bowel disease, immune colitis) that has required systemic treatment in the past 2 years. Replacement therapy (e.g.thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
   4. Known active CNS metastases and/or carcinomatous meningitis.

   i. Note: Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks before the first dose of study treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and have not required steroids for at least 7 days before study treatment. e. History of long QT syndrome or history or presence of an abnormal ECG that, in the Investigator's opinion, is clinically meaningful. Screening QTc interval > 450 milliseconds is excluded (corrected by Fridericia). In the event that a single QTc is > 450 milliseconds, the patient may enrol if the average QTc for the 3 ECGs is < 450 milliseconds. For patients with an intraventricular conduction delay (QRS interval > 120 msec), the JTc interval may be used in place of the QTc with Sponsor approval. The JTc must be < 340 milliseconds if JTc is used in place of the QTc. Patients with left bundle branch block are excluded.

   f. History of or current risk factor for torsade de pointes (e.g., heart failure, hypokalaemia, or a family history of long QT syndrome). g. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrolment), myocardial infarction (< 6 months prior to enrolment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or any of the following (<6 months prior to enrolment): acute coronary syndromes, coronary angioplasty or bypass grafting, serious cardiac arrhythmia requiring medication including second degree (Type 2) or third degree AV block, cardiomyopathy, pericarditis or myocarditis.

   h. Any history of interstitial lung disease or pneumonitis. i. History of allogenic stem cell transplantation or organ transplantation. j. Cirrhosis or current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, oesophageal/ gastric varices, persistent jaundice k. Women who are pregnant or breastfeeding l. Active infection requiring systemic therapy. m. Patients with active malignancy requiring concurrent intervention or previous malignancies (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colon, endometrial, cervical/dysplasia, melanoma or breast) unless a complete remission was achieved at least 2 years prior to study entry and no additional therapy is required during the study period.

   n. Any serious or uncontrolled medical disorder or active infection that, in the opinion of the Investigator, may increase the risk associated with study participation, study drug administration, or would impair the ability of the patient to receive protocol therapy.
5. Treatment with anticancer medications, investigational drugs, surgery and/or radiation within the following interval before the first administration of study drug:

   1. <90 days for prior taxane.
   2. <14 days for chemotherapy, targeted small-molecule therapy, surgical resection of lesions or radiation therapy (prior palliative radiotherapy must have been completed at least 14 days prior to study drug administration). Patients must also not require corticosteroids and must have recovered from pneumonitis as a result of treatment and show no evidence of pneumonitis for at least 1 month. A 1-week washout is permitted for palliative radiation to non-CNS disease with Sponsor approval. Note: The use of denosumab is permitted.
   3. < 14 days for a prior PD1 pathway-targeted agent.
   4. < 28 days for prior monoclonal antibody used for anticancer therapy with the exception of PD1 pathway-targeted agents.
   5. < 28 days or 5 half-lives (whichever is longer) before the first dose for all other investigational study drugs or devices. For investigational agents with long halflives (e.g., > 5 days), enrolment before the fifth half-life requires Medical Monitor approval.
   6. Radiotherapy -At least 6 weeks from prior radioisotope therapy. Note: Investigational agents that are not designed as antineoplastic treatment but used in combination with standard therapies are allowed.
6. Receiving an immune-suppressive based treatment for any reason (including chronic use of systemic corticosteroid at doses > 10 mg/day prednisone equivalent) within 14 days prior to the first dose of study treatment. Use of inhaled or topical steroids (including but not limited to creams or intra-articular injection) or brief corticosteroid use for radiographic procedures or systemic corticosteroids ≤ 10 mg is permitted.
7. Have received a live vaccine within 30 days of planned start of study therapy while on trial. With regards to other type of vaccines, including SARS-Co2 vaccines, are allowed.
8. Known allergy or reaction to any component of either study drugs or formulation components.
9. Known alcohol or other substance abuse.
10. Laboratory and medical history parameters not within Protocol-defined range. Cycle 1 Day 1 laboratory assessments for the determination of eligibility do not need to be performed if the screening laboratory assessments were performed within 7 days of Cycle 1 Day 1. If the screening laboratory assessments were performed more than 7 days before Cycle 1 Day 1, then the haematology and serum chemistry laboratory results must be confirmed up to 3 days before treatment initiation on Cycle 1 Day 1.

    1. Absolute neutrophil count < 1.5 × 109/L.
    2. Platelet count < 100 × 109/L.
    3. Haemoglobin < 9 g/dL (transfusion is acceptable to meet this criterion).
    4. Serum creatinine ≥ 1.5 × institutional upper limit of normal (ULN) or measured or calculated creatinine clearance (CrCl) (glomerular filtration rate can also be used in place of creatinine or CrCl) < 50 mL/min for patients with creatinine levels > 1.5 × institutional ULN.
    5. Aspartate aminotransferase (AST) or ALT ≥ 2.5 × ULN in the absence of hepatic metastases or ≥ 5 × ULN with hepatic metastases at screening.
    6. Total bilirubin ≥ 1.2 × ULN are excluded unless direct bilirubin is ≤ ULN. If there is no institutional ULN, then direct bilirubin must be < 40% of total bilirubin to be eligible (except patients with Gilbert syndrome, who must have total bilirubin < 51.3 μmol/L).
    7. International normalized ratio or prothrombin time (PT) > 1.5 × ULN.
    8. Activated partial thromboplastin time (aPTT) > 1.5 × ULN.
    9. Evidence of acute infection of hepatitis B virus (HBV), (for example: positive for HBsAg, anti-HBc, IgM anti-HBc and negative for anti-HBs), hepatitis C virus (HCV) (for example: HCV antibody reactive; HCV RNA detected) and Human Immunodeficiency Virus (HIV). Patients who are on stable antiviral therapy for their viral infection of hepatitis (e.g., HBV, HCV) or HIV (i.e., for at least 12 months) and willing to remain on these during and for 6 months after end of study treatment, and/or asymptomatic are eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE V5 | On Day 1 and Day 15 of Cycle 1; Day 1 of Cycle 2 onwards. Each cycle is 21 days
  Safety measured by AEs
To compare across treatment arms the proportion of patients with a reduction in peripheral blood Tregs (for example as defined by CD4+CD25+CD127- expression) | On Day 1 of each Cycle. Cycle length is 21 days
  Change from baseline of at least 50% by Day 42 as assessed by mass cytometry (cytometry by time of flight, CyTOF)
Number of Participants With changes in laboratory parameters | On Day 1and Day 15 of Cycle 1; Day 1 of Cycle 2 onwards. Each cycle is 21 days
  Measures by chemistry and haematology laboratory parameters
Number of Participants with Changes in ECG from baseline | On Day 1 and Day 15 of Cycle 1; Day 1 of Cycle 2 onwards. Each cycle is 21 days
  Measured by 12 Lead ECG
Number of Participants With Change on Physical Examination from Baseline | On Day 1and Day 15 of Cycle 1; Day 1 of Cycle 2 onwards. Each cycle is 21 days
  Measured by physical examination

SECONDARY OUTCOMES:
To further evaluate immune cell subsets in peripheral blood following treatment with roginolisib when given in combination with dostarlimab, and with/without docetaxel | On Day 1 of each cycle up to 36 weeks. Each cycle is 21 days
  Change from baseline in immune related signatures as assessed by mass cytometry (expanded analyses using the same sample used for the primary endpoint)
To evaluate preliminary signs of clinical efficacy of roginolisib when given in combination with dostarlimab, and with/without docetaxel | Every 6 weeks whilst on treatment anticipated to be 36 weeks
  Objective Response Rate (ORR) per RECIST v1.1 as assessed by the investigator
To evaluate preliminary signs of clinical efficacy of roginolisib when given in combination with dostarlimab, and with/without docetaxel | Every 6 weeks whilst on treatment anticipated to be 36 weeks
  Duration of response (DOR) per RECIST v1.1 as assessed by the investigator
To evaluate preliminary signs of clinical efficacy of roginolisib when given in combination with dostarlimab, and with/without docetaxel | Every 6 weeks whilst on treatment anticipated to be 36 weeks
  Disease Control Rate (DCR) per RECIST v1.1 as assessed by the investigator
To evaluate preliminary signs of clinical efficacy of roginolisib when given in combination with dostarlimab, and with/without docetaxel | Every 6 weeks whilst on treatment anticipated to be 36 weeks
  Clinical Benefit Rate (CBR) per RECIST v1.1 as assessed by the investigator
To evaluate preliminary signs of clinical efficacy of roginolisib when given in combination with dostarlimab, and with/without docetaxel | Every 6 weeks whilst on treatment anticipated to be 36 weeks
  Progression free survival (PFS) per RECIST v1.1 as assessed by the investigator
To evaluate preliminary signs of clinical efficacy of roginolisib when given in combination with dostarlimab, and with/without docetaxel | Every 12 weeks after safety follow-up until their death or end of study
  Overall survival (OS)
Pharmacokinetic (PK) concentration of roginolisib when given in combination with dostarlimab, and with/without docetaxel | Day 1 of each whilst on treatment anticipated to be 36 weeks. Cycle length is 21 days
  Plasma concentrations of roginolisib

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lahn, MD, Study Director — iOnctura
Locations (7):
- Belgium (2):
  - Antwerp University Hospital, Antwerp
  - AZ Delta VZW, Roeselare
- Italy (2):
  - Istituto Romagnolo per lo studio dei Tumori "Dino Amadori", Meldola, Forlì-Cesena
  - Humanitas University, Department of Medical Oncology, Rozzano, Milan
- Spain (3):
  - Institut Català d'Oncologia Hospitalet, Barcelona
  - Hospital Universitari Son Espases, Palma
  - Hospital Universitario y Politécnico La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Undecided